CLINICAL TRIAL: NCT04251624
Title: A Randomized Control Trial Examining the Treatment Efficacy of a Novel Approach to Cognitive Remediation in Public Safety Personnel With Post-traumatic Stress Disorder (PTSD) and Co-morbid Conditions
Brief Title: Investigating the Use of Goal Management Therapy in Improving Cognitive Functioning in Public Safety Personnel With PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Homewood Research Institute (Other)
Collaborators: McMaster University (Other); St. Joseph's Healthcare Hamilton (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Homewood Health Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-05
Record Dates: First submitted 2019-08-12; First posted 2020-02-05 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Post Traumatic Stress Disorder; Cognitive Deficit
Keywords: cognitive remediation; public safety personnel; psychosocial education; first responders; military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Cognition Disorders

STUDY DESIGN:
Intervention Model Description: Participants assigned to the experimental group (Goal Management Therapy) will receive either 6 (phase 1) or 9 (phase 2 and phase 3) group therapy sessions.
  The matched control group (psychosocial education) will receive an equal number of group therapy sessions.
  Each session will be 2 hours long.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal Management Therapy (Experimental): Goal Management Therapy is a structured, short-term, present-oriented cognitive remediation program with emphasis on mindfulness and practice in planning and completion of goal-oriented behaviors.
  The primary objective of GMT is to train patients to interrupt ongoing behavior through the resumption of executive control in order to define goal hierarchies and monitor performance in achieving goals. Sessions include instructional material, interactive tasks, discussion of patients' real-life deficits, and homework assignments.
  Phase 1: Inpatients will attend group sessions twice per week for 3 weeks, each session being 2 hours in length.
  Phase 2: Outpatients from the community will attend 1 session per week for 9 weeks, each session being 2 hours in length.
  Phase 3: Outpatients from the community will attend 1 session per week for 9 weeks, each session being 2 hours in length.
  Interventions: Behavioral: Goal Management Therapy
- Psychosocial Education (Active Comparator): Psychosocial education will provide participants with educational materials (e.g., brain function, neuroplasticity) and lifestyle interventions (e.g., sleep hygiene, stress, exercise).
  They will be matched for length and for amount of facilitator contact with the Goal Management Therapy sessions.
  Phase 1: Inpatients will attend group sessions twice per week for 3 weeks, each session being 2 hours in length.
  Phase 2: Outpatients from the community will attend 1 session per week for 9 weeks, each session being 2 hours in length.
  Phase 3: Outpatients from the community will attend 1 session per week for 9 weeks, each session being 2 hours in length.
  Interventions: Behavioral: Psychosocial Education

INTERVENTIONS:
Behavioral: Goal Management Therapy — A cognitive training program aimed at improving cognitive deficits such as in memory, attention, learning, and executive functioning.
  Other Names: Goal Management Training
  Arms: Goal Management Therapy
Behavioral: Psychosocial Education — A group therapy program focusing on brain function, neuroplasticity, and lifestyle interventions.
  Arms: Psychosocial Education

SUMMARY:
This study examines the efficacy of Goal Management Therapy (GMT) - a well-established cognitive remediation strategy aimed at improving goal-directed behaviors that are dependent on basic cognitive processes and on executive functioning - among public safety personnel with post-traumatic stress disorder.

DETAILED DESCRIPTION:
Goal Management Therapy is a structured, short-term, CBT-based, cognitive remediation program with an emphasis on mindfulness, and practice in planning and completion of goal-oriented behaviours. The primary objective of GMT is to train participants to interrupt ongoing, disruptive behaviour through the resumption of executive control, in order to define goal hierarchies and monitor performance in achieving goals. Sessions include instructional material, interactive tasks, discussion of real-life deficits, and homework/practice activities.

The matched psychosocial education control group will focus on educating participants on topics like brain function and neuroplasticity, and on practicing lifestyle interventions (e.g., sleep hygiene, stress management, exercise).

The study will take place in three phases:

Phase 1 will consist of 6 sessions of Goal Management Therapy and 6 sessions of psychosocial education among public safety personnel and civilians who are inpatients at a mental health and addiction facility.

Phase 2 will consist of 9 sessions of Goal Management Therapy and 9 sessions of psychosocial education among public safety personnel who are members of the local community.

Phase 3 will consist of 9 sessions of Goal Management Therapy and 9 sessions of psychosocial education among public safety personnel who are members of the local community. This phase will also use functional Magnetic Resonance Imaging (fMRI) scans to investigate potential changes in the neurobiology of participants' brains.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of post-traumatic stress disorder on the Clinician Administered PTSD Scale (CAPS)
* are able to provide written informed consent

Exclusion Criteria:

* receiving treatment with anti-cholinergics, anti-psychotic medication, or psychostimulants
* use of benzodiazepines within the last 24 hours
* have had Electroconvulsive therapy within the past year
* a diagnosis of substance dependence or abuse within the past 6 months
* a recent history (within the past 12 months) of medical disorder known to adversely affect cognition
* a history of head trauma with more than one minute of loss of consciousness or a history of traumatic brain injury
* a history of neurological disorder
* a diagnosis of psychotic disorder or bipolar disorder
* a history of a neurodevelopmental disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in Score on the Delis-Kaplan Executive Function System (D-KEFS) Tower Test | Phase 1 (inpatient): Baseline and post-intervention at 3 weeks
  A neuropsychological assessment of planning, rule learning, response inhibition, and perseveration. Six scores are calculated: i) Total Achievement Score, which is the sum of achievement scores for all items administered. ii) Mean First-Move Time which reflects the average of the examinee's first move times. iii) Time-Per-Move Ratio, which indicates the average time the examinee takes to make each of his or her moves. iv) Move Accuracy Ratio is a means of assessing the efficiency with which the examinee constructed the towers. v) Total Rule Violations represents the total number of rule violations committed by the examinee across all items administered. vi) Rule-Violations-Per Item Ratio, reflects the average number of rule violations made by the examinee relative to the number of items administered. The total number of rule violations across all items administered is divided by the number of items administered. Higher scores indicate greater executive functioning performance.
Change in Score on the Wechsler Adult Intelligence Scale-IV (WAIS-IV) Coding subtest | Phase 1 (inpatient): Baseline and post-intervention at 3 weeks
  A neuropsychological assessment of processing speed. In a time limit of 120 seconds, the participant copies symbols that are paired with numbers based on a symbol key. The total raw score is calculated by scoring 1 point for each correctly drawn symbol completed within the time limit. Raw scores range between 0 and 135 points. The raw score is converted to a scaled score corrected for age and the scaled score may range between 1 and 19. Higher scaled scores indicate greater processing speed than lower scaled scores.
Change in Score on Conners Continuous Performance Task Third Edition (CPT-3) | Phase 1 (inpatient): Baseline and post-intervention at 3 weeks
  A neuropsychological assessment of inattentiveness, impulsivity, sustained attention, and vigilance. Values include:
  i) D-prime-discrimination of non targets from targets; ii) Omissions- all missed targets; iii) Commissions- all incorrect responses to non-targets; iv) Perseverations- response in less than 100 milliseconds following the presentation of a stimulus; v) Hit Reaction Time- mean response speed measured in milliseconds for all non-perseverative responses made during the entire administration; vi) Hit Reaction Time SD-consistency of response speed to targets for the entire administration; vii) Variability- response speed consistency; viii) Hit Reaction Time Block Change- slope of change in Hit Reaction Time across the six blocks of the administration; and ix) Hit Reaction Time Inter-Stimulus Interval Change slope of change in reaction time across the three inter-stimulus intervals. All scores are presented in T scores with higher T scores indicating worse performance.
Change in Score on the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Phase 1 (inpatient): Baseline, post-intervention at 3 weeks, and post-intervention at 3 months
  The WHODAS 2.0 is a 12-item self-report measure of six functional domains, including cognition, mobility, self-care, getting along with others, life activities, and participation in the community. The WHODAS 2.0 uses a Likert scale ranging from 0 ("No difficulty") to 4 ("Extreme difficulty or cannot do"). Values across the 12 items are summed, with the total score ranging between 0 and 48. Higher values indicate greater functional impairment.
Change from Baseline in Score on the Cognitive Failures Questionnaire (CFQ) at 3 weeks post-intervention and 3 months post-intervention | Phase 1 (inpatient): Baseline, post-intervention at 3 weeks, and post-intervention at 3 months. This measure will also be administered during week 1, week 3, week 6, and week 9 of the intervention.
  The CFQ is a 25-item self-report measure that captures daily errors in distractibility, blunders, names, and memory. Each item is rated on a Likert scale from 0 ("Never") to 4 ("Very often"). The CFQ has four subscales that include: i) Memory (i.e., sum of scores on items 16, 18, 12, 17, 23, 13, 6, 3 for a total score between 0 and 32); ii) Distractibility (i.e., sum of scores on items 1, 15, 2, 19, 21, 22, 3, 4, 25 for a total score between 0 and 36); iii) Blunders (i.e., sum of scores on items 9, 8, 10, 24, 5, 14, 11 for a total score between 0 and 28); and iv) Names (i.e., sum of scores on items 20 and 7 for a total score between 0 and 8). The CFQ total score is the sum of the 25 items, with total values ranging between 0 and 100. Higher scores indicate greater self-reported impairment in cognitive functioning.
Change in Score on the Return to Work Obstacles and Self-Efficacy Scale - Common Mental Disorders (ROSES-CMD) | Phase 1 (inpatient): Baseline and post-intervention at 3 weeks
  A 46-item questionnaire that assesses readiness to return to work in individuals with common mental disorders on 10 possible dimensions: fears of a relapse, cognitive difficulties, medication-related difficulties, job demands, feeling of organization injustice, difficult relation-immediate supervisor, difficult relations-co-workers, difficult relations-insurance company, difficult work/life balance, and loss of motivation to return to work. Items use a 7-point response scale and include specific questions to assess perceived obstacles (1=not an obstacle, 7=Big obstacle) and self-efficacy beliefs about overcoming the obstacles (1=not at all capable, 7=completely capable). Higher scores on 'obstacles' items and lower scores on 'self-efficacy' items indicate decreased readiness to return-to-work.
Change from Baseline in Score on the VOT Hooper Visual Organization Test at 3 weeks post-intervention | Phase 1 (inpatient): Baseline and post-intervention at 3 weeks
  A neuropsychological assessment of visual integration, the VOT requires individuals to identify common object that have been fragmented by mentally rearranging fragments of the object presented on a card, with a total of 30 cards. The VOT is scored by hand to obtain a single raw score, which is then corrected based on age and level of education. The corrected raw score is used to derive a T score, which is the value of interest. Higher T scores reflect better performance.
Change in Score on the Rey-Osterrieth Complex Figure Test (RCFT) | Phase 1 (inpatient): Baseline and post-intervention at 3 weeks
  A neuropsychological test in which participants are required to copy a complex drawing to provide insight into individuals visuospatial/visuoconstructive abilities and areas of executive functioning (e.g., planning, organization). A single raw score is computed by hand using a manualized procedure which is then converted to a T score. This computed T score is the value of interest for this study, with higher T scores reflecting better performance.
Change in Score on the Depression Anxiety Stress Scale (DASS-21) | Phase 1 (Inpatient): Week 1, Week 3, and Week 6 of intervention, and post-intervention at 3 weeks
  The DASS-21 is a self-report measure that assesses the presence and severity of symptoms of depression, anxiety, and stress over the last week. Respondents rate their symptoms on a 4-point scale with 0 representing absence of the symptom and 3 representing a symptom occurring almost all the time. Three scores are computed, one for each subscale (depression, anxiety, and stress), by summing all the values of the items on each respective subscale.
  The total scores for each subscale are then multiplied by 2. Higher scores reflect greater symptom severity and the calculated scores can be used to qualify the severity of the symptoms (e.g., normal/minimal, mild, moderate, severe, extremely severe).
Change in Score on the Stroop Colour and Word Test (SCWT) | Phase 1 (inpatient): Baseline and post-intervention at 3 weeks
  A neuropsychological test where individuals read colour words or names ink colors from different pages as quickly as possible within a time limit. It provides indices of processing speed and areas of executive functioning, such as cognitive flexibility, resistance to interference, and response inhibition. The test includes three stimulus sheets that yield three raw scores that are the number of words or ink colors read within the time limit (min = 0; no max score). Raw scores are converted to T scores using manualized procedures. Higher T scores indicate better performance.
Advanced Clinical Solutions Test of Premorbid Functioning (TOPF) | Phase 1 (inpatient): Baseline only
  The TOPF is a word-reading neuropsychological test that estimates an individual's level of cognitive and memory functioning before the onset of injury or illness. The test yields one raw score (total number of words correctly read before the discontinue criteria was met) that is converted to a T score. Higher T scores indicate better performance.
Change from baseline in scores on the PTSD Checklist for DSM-5 (PCL-5) at post-intervention | Phase 2 (outpatient): Baseline, week 3 of intervention, week 6 of intervention, post-intervention at 9 weeks, 3 months post-intervention, and 6 months post-intervention
  A 20-item self-report measure that assesses the severity of PTSD symptoms according to the diagnostic criteria outlined in the DSM-5. Symptom domains are intrusions, avoidance, negative alterations in mood and cognitions, and alterations in arousal and reactivity.
Change from baseline in scores on the Depression and Anxiety Stress Scale (DASS-21) at post-intervention | Phase 2 (outpatient): Baseline, week 3 of intervention, week 6 of intervention, post-intervention at 9 weeks, 3 months post-intervention, and 6 months post-intervention
  A self-report measure that assesses the presence and severity of symptoms of depression, anxiety, and stress over the last week. Respondents rate their symptoms on a 4-point scale with 0 representing absence of the symptom and 3 representing a symptom occurring almost all the time.
  Three scores are computed, one for each subscale (depression, anxiety, and stress), by summing all the values of the items on each respective subscale.
Change from baseline in scores on the Sustained Attention Response Task (SART) | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  Assesses sustained attention by requiring participants to withhold behavioural response to a single, infrequent target presented among a background of frequent non-targets; administered using Inquisit Web by Millisecond (software for administering neuropsychological testing online).
Change from baseline in scores on the Cognitive Failures Questionnaire (CFQ) at post-intervention | Phase 2 (outpatient): Baseline, week 3 of intervention, week 6 of intervention, post-intervention at 9 weeks, 3 months post-intervention, and 6 months post-intervention
  A 25-item measure of self-reported cognitive impairment that captures daily errors in distractibility, blunders, names, and memory. Each item is rated on a Likert scale from 0 ("Never") to 4 ("Very often").
Change from baseline in symptom severity as assessed by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  A 30-item structured, clinician-administered interview used to make a lifetime or current diagnosis of PTSD and to assess PTSD symptoms. Questions target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms on social and occupational functioning, and specifications for the dissociative subtype.
Functional neurological change from baseline at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  Functional Magnetic Resonance Imaging (fMRI) scans done at baseline and post-intervention will be compared to determine whether changes are apparent, post-intervention, in the functional organisation of the Central Executive Network (CEN)
Functional neurological change from baseline at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  Functional Magnetic Resonance Imaging (fMRI) scans done at baseline and post-intervention will be compared to determine whether changes are apparent, post-intervention, in myelin amounts in regions associated with cognitive function
Change from baseline in score on the Sustained Attention Response Task (SART) adapted for functional Magnetic Resonance Imaging (fMRI) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  A computer-based 'Go/No-Go' task adapted for fMRI that requires participants to inhibit a behavioural response to a single, infrequent target appearing amidst a presentation of frequent non-targets.
  Participants will be asked to press a button for every number presented except "3", under two conditions:
  1. a randomized presentation of numbers in two sets, each lasting one minute, and,
  2. a sequential presentation of numbers. Each condition will be presented three times. The second presentation of the numbers will be preceded by certain specific emotion-evoking 'trauma words' identified by the participant at a prior appointment.

SECONDARY OUTCOMES:
Demographic Information | Phase 1 (inpatient): administered at baseline only
  Self-report of demographic information, including age, sex, race, education, marital status, employment status, and employment type (e.g., active military member, veteran, public safety personnel, first responder, or other).
Mini International Neuropsychiatric Interview 7.0 (M.I.N.I.) | Phase 1 (inpatient): administered at baseline only
  The M.I.N.I. is a structured clinician administered interview to assess psychiatric disorders according to the Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5).
  The M.I.N.I. is divided into modules identified by letters, each corresponding to a diagnostic module. At the end of each module, diagnostic boxes permit the clinician to indicate whether diagnostic criteria are met. The diagnostic modules utilized within the study include:
  i) Major Depressive Episode
  ii) Suicidality
  iii) Manic and Hypomanic Episodes
  iv) Panic Disorder
  v) Agoraphobia
  vi) Social Anxiety Disorder
  vii) Obsessive Compulsive Disorder
  viii) Alcohol Use Disorder
  ix) Substance Use Disorder
  x) Psychotic Disorders and Mood Disorder with Psychotic Features
  xi) Anorexia Nervosa
  xii) Bulimia Nervosa
  xiii) Binge Eating Disorder; and
  xiiii) Generalized Anxiety Disorder.
Change in score on the PTSD Checklist for DSM-5 (PCL-5) | Phase 1 (inpatient): administered at 3 months post-intervention. This measure will also be administered during week 1, week 3, week 6, and week 9 of the intervention.
  The PCL-5 is a 20-item self-report measure that assesses the severity of PTSD symptoms according to the diagnostic criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5).
  The symptom domains are:
  intrusions (items 1 through 5; scores summed for a total between 0 and 20),
  avoidance (items 6 through 7; scores summed for a total between 0 and 8),
  negative alterations in mood and cognitions (items 8 through 14; scores summed for a total between 0 and 28), and
  alterations in arousal and reactivity (items 15 through 20; scores summed for a total between 0 and 24).
  Participants rate the severity of their symptoms in the past month on a Likert scale from 0 ("Not at all") to 4 ("Extremely"). A total PCL-5 score is derived by summing all the values of the items and the total score may range between 0 and 80.
  A cut-off point of 33 is suggested to indicate a probable PTSD diagnosis.
Change in Score on the Multiscale Dissociation Inventory (MDI) | Phase 1 (inpatient): administered during week 1, week 3, week 6, and week 9 of the intervention and at 3 months post-intervention
  The MDI is a 30-item self-report measure that assesses six domains of dissociative symptoms over the past month:
  disengagement (items 1, 7, 13, 19, 25; scores summed for a total between 5 and 25),
  depersonalization (items 2, 8, 14, 20, 26; scores summed for a total between 5 and 25),
  derealization (items 3, 9, 15, 21, 27; scores summed for a total between 5 and 25),
  emotional constriction (items 4, 10, 16, 22, 28; scores summed for a total between 5 and 35),
  memory disturbance (items 5, 11,17,23,29; scores summed for a total between 5 and 25), and
  identity dissociation (items 6, 12, 18, 24, 30; scores summed for a total between 5 and 25).
  Participants rate the severity of their symptoms within the last month on a Likert scale from 1 ("Never") to 5 ("Very often"). A total MDI score is derived by summing all the values of the items and the total score may range between 30 and 150.
  Higher total scores indicate greater dissociation.
Change in accuracy of episodic memory recall as measured using a standard EEG | Phase 1 (inpatient): baseline, post-intervention at 3 weeks.
  The standard EEG is performed using a 16 channel dry electrode wireless EEG headset designed to study the dynamics of large-scale brain networks known to impact mood, cognition, and behavior.
  Participants will be presenting with a total of 10 alternating blocks of autobiographical memory and working memory trials. They will be asked to describe 10 positive or neutral specific event memories in vivid detail. Additionally, they will be asked to identify 10-15 words/ phrases that would uniquely elicit these memories.
  They will then imagine themselves in 10 future imagined events, with 10-15 words/phrases that would uniquely elicit these imagined memories.
Demographic Information | Phase 2 (outpatient): collected at baseline only
  Age, sex, race, education, marital status, employment status, and employment type (e.g., active military member, veteran, public safety personnel, first responder, or other).
Change from baseline in scores on the Multiscale Dissociation Inventory (MDI) at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  A 30-item self-report measure that assesses six domains of dissociative symptoms over the past month -- disengagement, depersonalization, derealization, emotional constriction, memory disturbance, and identity dissociation.
Change from baseline in scores on the Difficulties in Emotion Regulation Scale (DERS) at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  A 36-item self-report measure that assesses difficulties with emotion regulation across six domains -- nonacceptance of emotional responses, difficulty engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity.
Change from baseline in scores on the Toronto Alexithymia Scale (TAS) at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  A 20-item self-report measure that assesses difficulties recognizing and naming emotions across three domains -- difficulty identifying feelings, difficulty describing feelings, and externally oriented thinking.
Change from baseline in scores on selected subtests of the CBS Research battery at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  The Double Trouble, Feature Match, Spatial Planning, and Odd One Out subtests of the CBS Research Battery will be administered remotely using Cambridge Brain Sciences (CBS; a web-based platform for assessing cognitive functioning), and Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess executive functioning, processing speed, and attention.
Change from baseline in scores on Digit Symbol Substitution Task at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  Digit Symbol Substitution Task will be administered remotely using Inquisit Web by Millisecond (software for administering neuropsychological testing online) to assess processing speed and attention.
Change from baseline in scores on selected subtests of the CBS Research battery at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  The Paired Associates and Digit Span subtests of the CBS Research Battery will be administered remotely using Cambridge Brain Sciences (CBS; a web-based platform for assessing cognitive functioning) and Zoom for healthcare (a PHIPA-compliant video conferencing platform) to assess declarative memory.
Change from baseline in scores on the Hopkins Verbal Learning Test-Revised (HVLT-R) at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  The Hopkins Verbal Learning Test-Revised (HVLT-R) will be administered remotely using Zoom for healthcare (a PHIPA-compliant video conferencing platform) to assess declarative memory.
Change from baseline in scores on selected subtests of the CBS Research battery at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  The Grammatical Reasoning subtest of the CBS Research Battery will be administered remotely using Cambridge Brain Sciences (CBS; a web-based platform for assessing cognitive functioning), and Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess the ability to quickly understand and make valid conclusions about concepts expressed in words.
Change from baseline in scores on selected subtests of the CBS Research battery at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  The Rotations and Polygons subtests of the CBS Research Battery will be administered remotely using Cambridge Brain Sciences (CBS; a web-based platform for assessing cognitive functioning) Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess visuospatial/visuoconstructive ability and sensorimotor integration.
Change from baseline in scores on the Rey Complex Figure Task (RCFT) at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  The Rey Complex Figure Task (RCFT) will be administered remotely using Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess visuospatial/visuoconstructive ability and sensorimotor integration.
Change from baseline in scores on selected subtests of the CBS Research battery at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  The Token Search, Monkey Ladder, and Spatial Span subtests of the CBS Research Battery will be administered remotely using Cambridge Brain Sciences (CBS; a web-based platform for assessing cognitive functioning) and Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess visual and visuospatial working memory.
Change from baseline in scores on the Return to work Obstacles and Coping Efficacy - Common Mental Disorders (ROSES-CMD) at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  Evaluates obstacles participants may face when returning to work (part A) and how capable they feel they are of overcoming them (part B).
  Items use a 7-point response scale and include specific questions to assess perceived obstacles and self-efficacy beliefs about overcoming the obstacles.
  Higher scores on 'obstacles' items and lower scores on 'self-efficacy' items indicate decreased readiness to return-to-work.
Change from baseline in scores on the World Health Organization's Disability Assessment Schedule (WHODAS 2.0) at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  A self-report measure that assesses health and disability on six domains of functioning in life: cognition, mobility, self-care, getting along (interacting with others), life activities, and participation (participating in society).
Change from baseline in scores on the Lam Employment Absence and Productivity Scale (LEAPS) at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  A self-report measure designed to assess and monitor work functioning and productivity. Participants are asked to respond to 4 questions; the fourth question assesses specific symptoms by having participants respond to 7 sub-questions on a 5-point scale.
  Two values of interest for this study are derived:
  i) measure of work impairment (sum of responses to the 7 sub-questions) ii) percent of work hours missed due to impairment [raw score of item 3 (hours of work missed) divided by raw score of item 2 (hours of work scheduled) multiplied by 100.
Change from baseline in scores on the Sheehan Disability Scale (SDS) at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  A 3-item self-report measure of disability in work, social relationships, and family life. Items are scored on a Likert scale between 0 and 10 and are summed into a single dimensional measure of global functional impairment.
  Total score may range from 0 to 30, with higher scores indicating greater impairment.
Change from baseline in scores on the BADS Dysexecutive Questionnaire (DEX) at post-intervention | Phase 2 (outpatient): Baseline, post-intervention at 9 weeks, 3 months post-intervention, 6 months post-intervention
  A 20-item measure of self-reported cognitive impairment that asks participants to rate inhibition, positive and negative affect, memory, and intention. Each item is rated on a Likert scale from 0 ("Never") to 4 ("Very often").
Scores on the Life Events Checklist for DSM-5 (LEC-5) at baseline | Phase 2 (outpatient): Administered at baseline only
  A self-report measure designed to screen for potentially traumatic events in a respondent's lifetime by assessing exposure to 16 events known to potentially result in PTSD or distress, as well as one additional item to assess any other extraordinarily stressful event not captured in the first 16 items.
Scores on the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) at baseline | Phase 2 (outpatient): Administered at baseline only
  A 30-item structured, clinician-administered interview used to make a lifetime or current diagnosis of PTSD and to assess PTSD symptoms. Questions target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms on social and occupational functioning, and specifications for the dissociative subtype.
Scores on the Mini International Neuropsychiatric Interview (M.I.N.I.) 7.0 at baseline | Phase 2 (outpatient): Administered at baseline only
  A structured clinician-administered interview that assesses psychiatric disorders according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition.
  Diagnostic modules utilized within the study include i) Major Depressive Episode; ii) Suicidality; iii) Manic and Hypomanic Episodes; iv) Panic Disorder; v) Agoraphobia; vi) Social Anxiety Disorder; vii) Obsessive Compulsive Disorder; viii) Alcohol Use Disorder; ix) Substance Use Disorder; x) Psychotic Disorders and Mood Disorder with Psychotic Features; xi) Anorexia Nervosa; xii) Bulimia Nervosa; xiii) Binge Eating Disorder; and xiiii) Generalized Anxiety Disorder.
Scores on the Moral Injury Events Scale (MIES) at baseline | Phase 2 (outpatient): Administered at baseline only
  A 9-item self-report measure assessing moral injury along two dimensions in military and veteran populations -- perceived transgressions and perceived betrayals.
Scores on the Childhood Trauma Questionnaire (CTQ) at baseline | Phase 2 (outpatient): Administered at baseline only
  A self-report measure that assesses for exposure to five forms of common childhood trauma -- sexual abuse, physical abuse, emotional abuse, physical neglect, emotional neglect.
Scores on the Advanced Clinical Solutions (ACS) Test of Premorbid Functioning (TOPF) at baseline | Phase 2 (outpatient): Administered at baseline only
  The Advanced Clinical Solutions (ACS) Test of Premorbid Functioning (TOPF) provides an estimate of pre-morbid intellectual functioning, and will be administered using Zoom for Healthcare (a PHIPA-compliant video conferencing platform).
Demographic Information | Phase 3 (fMRI): Collected at baseline only
  Age, sex, race, education, relationship status, employment status, and profession (whether police, firefighter, volunteer firefighter, search and rescue personnel, paramedic, nurse, correctional officer, probation officer, parole officer, or emergency dispatcher)
Change from baseline in scores on the Coding subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  The Coding subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) will be administered in-person to assess processing speed and attention.
Change from baseline in scores on the Symbol Search subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  The Symbol Search subtests of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) will be administered in-person to assess processing speed and attention.
Change from baseline in scores on selected subtests of the Creyos battery at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  The Double Trouble, Feature Match, Spatial Planning, and Odd One Out subtests of the Creyos battery will be administered remotely using Creyos (formerly known as CBS; a web-based platform for assessing cognitive functioning) and Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess executive functioning, processing speed, and attention.
Change from baseline in scores on the Digit Span subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  The Digit Span subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) will be administered in-person to assess declarative memory.
Change from baseline in scores on California Verbal Learning Test (CVLT-3) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  The California Verbal Learning Test (CVLT-3, standard and alternate forms) will be administered over Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess declarative memory.
Change from baseline in scores on selected subtests of the Creyos battery at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  The Paired Associates and Digit Span subtests of the Creyos battery will be administered remotely using Creyos (formerly known as CBS; a web-based platform for assessing cognitive functioning) and Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess declarative memory.
Change from baseline in scores on selected subtests of the Creyos battery at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  The Grammatical Reasoning subtest of the Creyos Battery will be administered remotely using Creyos (formerly known as CBS; a web-based platform for assessing cognitive functioning) and Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess the ability to quickly understand and make valid conclusions about concepts expressed in words.
Change from baseline in scores on selected subtests of the Creyos battery at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  The Rotations and Polygons subtests of the Creyos Battery will be administered remotely using Creyos (formerly known as CBS; a web-based platform for assessing cognitive functioning) and Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess visuospatial/visuoconstructive ability and sensorimotor integration.
Change from baseline in scores on selected subtests of the Creyos battery at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  Token Search, Monkey Ladder, and Spatial Span subtests of the CBS Research Battery will be administered remotely using Creyos (formerly known as CBS; a web-based platform for assessing cognitive functioning) and Zoom for Healthcare (a PHIPA-compliant video conferencing platform) to assess visual/visuospatial working memory.
Change from baseline in score on the Depression and Anxiety Stress Scale (DASS-21) at post-intervention | Phase 3 (fMRI): Baseline, week 3 of intervention, week 6 of intervention, and post-intervention at 9 weeks
  A self-report measure that assesses the presence and severity of symptoms of depression, anxiety, and stress over the last week. Respondents rate their symptoms on a 4-point scale with 0 representing absence of the symptom and 3 representing a symptom occurring almost all the time. Three scores are computed, one for each subscale (depression, anxiety, and stress), by summing all the values of the items on each respective subscale.
Change from baseline in score on the PTSD Checklist for DSM-5 (PCL-5) at post-intervention | Phase 3 (fMRI): Baseline, week 3 of intervention, week 6 of intervention, and post-intervention at 9 weeks
  A 20-item self-report measure that assesses the severity of PTSD symptoms according to the diagnostic criteria outlined in the DSM-5. Symptom domains are intrusions, avoidance, negative alterations in mood and cognitions, and alterations in arousal and reactivity.
Change from baseline in score on the Multiscale Dissociation Inventory (MDI) at post-intervention | Phase 3 (fMRI): Baseline, week 3 of intervention, week 6 of intervention, and post-intervention at 9 weeks
  A 30-item self-report measure that assesses six domains of dissociative symptoms over the past month -- disengagement, depersonalization, derealization, emotional constriction, memory disturbance, and identity dissociation.
Change from baseline in score on the Difficulties in Emotion Regulation Scale (DERS) at post-intervention | Phase 3 (fMRI): Baseline, week 3 of intervention, week 6 of intervention, and post-intervention at 9 weeks
  A 36-item self-report measure that assesses difficulties with emotion regulation across six domains -- nonacceptance of emotional responses, difficulty engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity.
Change from baseline in score on the Toronto Alexithymia Scale (TAS) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  A 20-item self-report measure that assesses difficulties recognizing and naming emotions across three domains -- difficulty identifying feelings, difficulty describing feelings, and externally oriented thinking.
Change from baseline in score on the Moral Injury Assessment for Public Safety Personnel (MIA-PSP) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  A 17-item self-report measure of work-related morally injurious experiences unique to public safety personnel across three underlying factors -- perpetrations, betrayals, and emotional sequelae.
Change from baseline in scores on the BADS Dysexecutive Questionnaire (DEX) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  A 20-item measure of self-reported cognitive impairment that asks participants to rate inhibition, positive and negative affect, memory, and intention. Each item is rated on a Likert scale from 0 ("Never") to 4 ("Very often").
Change from baseline in scores on the Cognitive Failures Questionnaire (CFQ) at post-intervention | Phase 3 (fMRI): Baseline, week 3 of intervention, week 6 of intervention, and post-intervention at 9 weeks
  A 25-item measure of self-reported cognitive impairment that captures daily errors in distractibility, blunders, names, and memory. Each item is rated on a Likert scale from 0 ("Never") to 4 ("Very often").
Change from baseline in scores on the Return to work Obstacles and Coping Efficacy - Common Mental Disorders (ROSES-CMD) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  Evaluates obstacles participants may face when returning to work (part A) and how capable they feel they are of overcoming them (part B).
  Items use a 7-point response scale and include specific questions to assess perceived obstacles and self-efficacy beliefs about overcoming the obstacles.
  Higher scores on 'obstacles' items and lower scores on 'self-efficacy' items indicate decreased readiness to return-to-work.
Change from baseline in scores on the World Health Organization's Disability Assessment Schedule (WHODAS 2.0) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  A self-report measure that assesses health and disability on six domains of functioning in life: cognition, mobility, self-care, getting along (interacting with others), life activities, and participation (participating in society).
Change from baseline in scores on the Lam Employment Absence and Productivity Scale (LEAPS) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  A self-report measure designed to assess and monitor work functioning and productivity. Participants are asked to respond to 4 questions; the fourth question assesses specific symptoms by having participants respond to 7 sub-questions on a 5-point scale.
  Two values of interest for this study are derived:
  i) measure of work impairment (sum of responses to the 7 sub-questions) ii) percent of work hours missed due to impairment [raw score of item 3 (hours of work missed) divided by raw score of item 2 (hours of work scheduled) multiplied by 100.
Change from baseline in scores on the Sheehan Disability Scale (SDS) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  A 3-item self-report measure of disability in work, social relationships, and family life. Items are scored on a Likert scale between 0 and 10 and are summed into a single dimensional measure of global functional impairment.
  Total score may range from 0 to 30, with higher scores indicating greater impairment.
Change from baseline in scores on the Survey of Perceived Organizational Support (SPOS) at post-intervention | Phase 3 (fMRI): Baseline and post-intervention at 9 weeks
  Assesses the extent to which an individual believes that their organization is a) committed to them, b) values their continued membership, and c) is generally concerned about their well-being.
Scores on the Advanced Clinical Solutions (ACS) Test of Premorbid Functioning (TOPF) at baseline | Phase 3 (fMRI): Administered at baseline only
  The Advanced Clinical Solutions (ACS) Test of Premorbid Functioning (TOPF) provides an estimate of pre-morbid intellectual functioning, and will be administered using Zoom for Healthcare (a PHIPA-compliant video conferencing platform).
Scores on the Life Events Checklist for DSM-5 (LEC-5) at baseline | Phase 3 (fMRI): Administered at baseline only
  A self-report measure designed to screen for potentially traumatic events in a respondent's lifetime by assessing exposure to 16 events known to potentially result in PTSD or distress, as well as one additional item to assess any other extraordinarily stressful event not captured in the first 16 items.
Scores on the Mini International Neuropsychiatric Interview 7.0.2 (M.I.N.I.) at baseline | Phase 3 (fMRI): Administered at baseline only
  A structured clinician-administered interview that assesses psychiatric disorders according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition.
  Diagnostic modules utilized within the study include i) Major Depressive Episode; ii) Suicidality; iii) Manic and Hypomanic Episodes; iv) Panic Disorder; v) Agoraphobia; vi) Social Anxiety Disorder; vii) Obsessive Compulsive Disorder; viii) Alcohol Use Disorder; ix) Substance Use Disorder; x) Psychotic Disorders and Mood Disorder with Psychotic Features; xi) Anorexia Nervosa; xii) Bulimia Nervosa; xiii) Binge Eating Disorder; and xiiii) Generalized Anxiety Disorder.
Scores on the Childhood Trauma Questionnaire (CTQ) at baseline | Phase 3 (fMRI): Administered at baseline only
  A self-report measure that assesses for exposure to five forms of common childhood trauma -- sexual abuse, physical abuse, emotional abuse, physical neglect, emotional neglect.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McKinnon, PhD, Principal Investigator — McMaster University, St. Joseph's Healthcare Hamilton, Homewood Research Institute
Locations (1):
- Homewood Research Institute, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyd JE, Lanius RA, McKinnon MC. Mindfulness-based treatments for posttraumatic stress disorder: a review of the treatment literature and neurobiological evidence. J Psychiatry Neurosci. 2018 Jan;43(1):7-25. doi: 10.1503/jpn.170021. Epub 2017 Oct 2. PMID 29252162
- [Background] Boyd JE, Protopopescu A, O'Connor C, Neufeld RWJ, Jetly R, Hood HK, Lanius RA, McKinnon MC. Dissociative symptoms mediate the relation between PTSD symptoms and functional impairment in a sample of military members, veterans, and first responders with PTSD. Eur J Psychotraumatol. 2018 May 17;9(1):1463794. doi: 10.1080/20008198.2018.1463794. eCollection 2018. PMID 29805778
- [Background] McKinnon MC, Boyd JE, Frewen PA, Lanius UF, Jetly R, Richardson JD, Lanius RA. A review of the relation between dissociation, memory, executive functioning and social cognition in military members and civilians with neuropsychiatric conditions. Neuropsychologia. 2016 Sep;90:210-34. doi: 10.1016/j.neuropsychologia.2016.07.017. Epub 2016 Jul 18. PMID 27444881
- [Background] Meusel LA, Hall GB, Fougere P, McKinnon MC, MacQueen GM. Neural correlates of cognitive remediation in patients with mood disorders. Psychiatry Res. 2013 Nov 30;214(2):142-52. doi: 10.1016/j.pscychresns.2013.06.007. Epub 2013 Aug 30. PMID 23993991
- [Background] Lanius RA, Frewen PA, Tursich M, Jetly R, McKinnon MC. Restoring large-scale brain networks in PTSD and related disorders: a proposal for neuroscientifically-informed treatment interventions. Eur J Psychotraumatol. 2015 Mar 31;6:27313. doi: 10.3402/ejpt.v6.27313. eCollection 2015. PMID 25854674

DOCUMENTS (1):
  • Informed Consent Form (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT04251624/ICF_000.pdf